CLINICAL TRIAL: NCT02560363
Title: An Open-label, Randomized, Cross Over Single Oral Dose Study Comparing the Pharmacokinetics of Different Formulations of AZD9977 (Part A) and Influence of Food (Part B) in Healthy Male Subjects
Brief Title: A Study to Compare the Pharmacokinetics of Different Formulations of AZD9977 and the Influence of Food in Healthy Male Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Has been terminated before FSFV.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D6400C00003; 2015-002807-26 (EudraCT Number)
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Pharmacokinetics; Healthy Male Subjects; Safety; Food Effect
Keywords: AZD9977; Safety; Tolerability; Pharmacokinetics; Food effect; AZD9977 capsules; AZD9977 suspension
MeSH Terms: interventions — AZD9977; Suspensions; Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment sequence 1 (Experimental): Period 1:Fast ER formulation of AZD9977 Period 2:Intermediate ER formulation of AZD9977 Period 3:Slow ER formulation of AZD9977 Period 4:IR formulation of AZD9977 Period 5:Fast, intermediate or slow ER formulation with food
  Interventions: Drug: AZD9977 immediate release (IR) oral suspension; Drug: AZD9977 extended release (ER) capsules [fast]; Drug: AZD9977 extended release (ER) capsules [intermediate]; Drug: AZD9977 extended release (ER) capsules [slow]
- Treatment sequence 2 (Experimental): Period 1:Intermediate ER formulation of AZD9977 Period 2:IR formulation of AZD9977 Period 3:Fast ER formulation of AZD9977 Period 4:Slow ER formulation of AZD9977 Period 5:Fast, intermediate or slow ER formulation with food
  Interventions: Drug: AZD9977 immediate release (IR) oral suspension; Drug: AZD9977 extended release (ER) capsules [fast]; Drug: AZD9977 extended release (ER) capsules [intermediate]; Drug: AZD9977 extended release (ER) capsules [slow]
- Treatment sequence 3 (Experimental): Period 1:Slow ER formulation of AZD9977 Period 2:Fast ER formulation of AZD9977 Period 3:IR formulation of AZD9977 Period 4:Intermediate ER formulation of AZD9977 Period 5:Fast, intermediate or slow ER formulation with food
  Interventions: Drug: AZD9977 immediate release (IR) oral suspension; Drug: AZD9977 extended release (ER) capsules [fast]; Drug: AZD9977 extended release (ER) capsules [intermediate]; Drug: AZD9977 extended release (ER) capsules [slow]
- Treatment sequence 4 (Experimental): Period 1:IR formulation of AZD9977 Period 2:Slow ER formulation of AZD9977 Period 3:Intermediate ER formulation of AZD9977 Period 4:Fast ER formulation of AZD9977 Period 5:Fast, intermediate or slow ER formulation with food
  Interventions: Drug: AZD9977 immediate release (IR) oral suspension; Drug: AZD9977 extended release (ER) capsules [fast]; Drug: AZD9977 extended release (ER) capsules [intermediate]; Drug: AZD9977 extended release (ER) capsules [slow]

INTERVENTIONS:
Drug: AZD9977 immediate release (IR) oral suspension — 120 mg (4.8 mL x 25 mg/mL) oral suspension, single dose
Drug: AZD9977 extended release (ER) capsules [fast] — 120 mg (2 x 60mg capsules) single dose
Drug: AZD9977 extended release (ER) capsules [intermediate] — 120 mg (2 x 60mg capsules) single dose
Drug: AZD9977 extended release (ER) capsules [slow] — 120 mg (2 x 60mg capsules) single dose

SUMMARY:
This is an open-label, randomized, cross over single oral dose study to compare the pharmacokinetics of different formulations of AZD9977 in Part A and the influence of food in Part B in healthy male subjects

DETAILED DESCRIPTION:
This is an open-label, randomized, cross over single oral dose study to compare the pharmacokinetics of three different extended-release formulations and an immediate-release formulation (reference) of AZD9977 in Part A and the influence of food in Part B in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male subjects aged 18 to 50 years with suitable veins for cannulation or repeated venipuncture.
* Male subjects have to comply with the restrictions for sexual activity provided to them.
* Have a body mass index (BMI) between 18 and 32 kg/m2, inclusive, and weigh at least 50 kg.
* Subject judged likely to complete and agree to eat a specified high-fat, high-calorie standardized FDA breakfast.
* Able to understand, read and speak the English language.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
* Any clinically significant abnormalities in clinical chemistry, hematology or urinalysis results, as judged by the investigator.
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) antibody.
* Abnormal findings in vital signs, after 10 minutes resting in the supine position, defined as any of the following:

  * Systolic blood pressure (SBP) < 90 mmHg or ≥ 140 mmHg
  * Diastolic blood pressure (DBP) < 50 mmHg or ≥ 90 mmHg
  * Pulse < 45 or > 90 bpm
* Any clinically important abnormalities in rhythm, conduction or morphology of the electrocardiogram (ECG) at screening or pre-dose, as considered by the investigator.
* Prolonged QTcF > 450 ms or family history of long QT syndrome.
* PR (PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation).
* PR (PQ) interval prolongation > 240 ms; intermittent second (history of Wenckebach block while asleep is not exclusive) or third degree atrioventricular (AV) block or AV dissociation.
* Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB) or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of ventricular hypertrophy or pre-excitation.
* Serum potassium higher than 5.0 mmol/L at screening or admission to the study center (Day -1).
* Known or suspected history of drug abuse, as judged by the investigator.
* Current smokers or those who have smoked or used nicotine products within the 3 months prior to screening.
* History of alcohol abuse or excessive intake of alcohol as judged by the investigator.
* Positive screen for drugs of abuse, alcohol or cotinine at screening or admission to the study center.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD9977.
* Excessive intake of caffeine containing drinks or food (e.g., coffee, tea and chocolate) as judged by the investigator.
* Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to first dose of AZD9977.
* Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during 2 weeks prior to 1st dosing in Part A, or longer if the medication has a long half-life.
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest.
* Subjects who have previously received AZD9977
* Involvement of any AstraZeneca, PAREXEL, or study site employee or their close relatives.
* Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
* Subjects who are vegans, vegetarians or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the investigator.
* Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Rate and extent of absorption of the extended-release formulations in comparison with an immediate-release formulation of AZD9977 by assessment of Frel (AUC) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36 and 48 hours post-dose on each dosing day
  Relative bioavailability (Frel [AUC]) by assessement of the ratio of AUC (Area under plasma concentration-time curve from time zero extrapolated to infinity) between the extended-release formulations in comparison with an immediate-release formulation of AZD9977
Rate and extent of absorption of the extended-release formulations in comparison with an immediate-release formulation of AZD9977 by assessment of Frel (AUC0-t) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36 and 48 hours post-dose on each dosing day
  Relative bioavailability (Frel [AUC0-t]) by assessement of the ratio of AUC (Area under the plasma concentration-curve from time zero to time of last quantifiable concentration) between the extended-release formulations in comparison with an immediate-release formulation of AZD9977
Rate and extent of absorption of the extended-release formulations in comparison with an immediate-release formulation of AZD9977 by assessment of Frel (AUC0-24) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36 and 48 hours post-dose on each dosing day
  Relative bioavailability (Frel [AUC0-24]) by assessement of the ratio of AUC (Area under the plasma concentration-time curve from time zero to 24 hours post-dose) between the extended-release formulations in comparison with an immediate-release formulation of AZD9977
Rate and extent of absorption of the extended-release formulations in comparison with an immediate-release formulation of AZD9977 by assessment of Frel (Cmax) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36 and 48 hours post-dose on each dosing day
  Relative bioavailability (Frel [Cmax]) by assessement of the ratio of AUC (Observed maximum plasma concentration) between the extended-release formulations in comparison with an immediate-release formulation of AZD9977
Rate and extent of absorption of an extended-release formulation of AZD9977 under fasting condtions in comparision with fed condtions by assessment of Frel (AUC) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36 and 48 hours post-dose on each dosing day
  Relative bioavailability (Frel [AUC]) by assessement of the ratio of AUC (Area under plasma concentration-time curve from time zero extrapolated to infinity) after dosing of an extended-release formulation under fed and fasting conditions
Rate and extent of absorption of an extended-release formulation of AZD9977 under fasting condtions in comparision with fed condtions by assessment of Frel(AUC0-t) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36 and 48 hours post-dose on each dosing day
  Relative bioavailability (Frel [AUC0-t]) by assessement of the ratio of AUC (Area under the plasma concentration-curve from time zero to time of last quantifiable concentration) after dosing of an extended-release formulation under fed and fasting conditions
Rate and extent of absorption of an extended-release formulation of AZD9977 under fasting condtions in comparision with fed condtions by assessment of Frel(AUC0-24) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36 and 48 hours post-dose on each dosing day
  Relative bioavailability (Frel [AUC0-24]) by assessement of the ratio of AUC (Area under the plasma concentration-time curve from time zero to 24 hours post-dose) after dosing of an extended-release formulation under fed and fasting conditions
Rate and extent of absorption of an extended-release formulation of AZD9977 under fasting condtions in comparision with fed condtions by assessment of Frel(Cmax) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36 and 48 hours post-dose on each dosing day
  Relative bioavailability (Frel[Cmax]) by assessement of the ratio of AUC (Area under the plasma concentration-time curve from time zero to 24 hours post-dose) after dosing of an extended-release formulation under fed and fasting conditions

SECONDARY OUTCOMES:
Safety and tolerabilty of AZD9977 by assessment of the number of adverse events and the number of subjects with adverse events | From screening to post-study visit, up to 10 weeks
  To assess the safety and tolerability of single doses of AZD9977
Safety and tolerabilty of AZD9977 by assessment of cardiac telemetry | On Day -1 and pre-dose until 24 hours post dose on Day 1
  To assess the safety and tolerability of single doses of AZD9977
Safety and tolerabilty of AZD9977 by assessment of blood pressure | From screening to post-study visit, up to 10 weeks
  To assess the safety and tolerability of single doses of AZD9977
Safety and tolerabilty of AZD9977 by assessment of pulse | From screening to post-study visit, up to 10 weeks
  To assess the safety and tolerability of single doses of AZD9977
Safety and tolerability of AZD9977 by assessment of electrocardiogram | From screening to post-study visit, up to 10 weeks
  To assess the safety and tolerability of single doses of AZD9977
Safety and tolerability of AZD9977 by assessment of physical examination | From screening to post-study visit, up to 10 weeks
  This is a composite of the general appearance, skin, cardiovascular, respiratory, abdomen, head and neck (including ears, eyes, nose and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Safety and tolerability of AZD9977 by assessment of safety laboratory tests | From screening to post-study visit, up to 10 weeks
  This is a composite of clinical chemistry, hematology and urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MBChB, MSc, MFPM, Principal Investigator — Parexel
Locations (1):
- Research Site, Harrow, United Kingdom